CLINICAL TRIAL: NCT06380543
Title: Efficacy of ERCP Using ESGE Algorithm for Biliary Cannulation: a Multicenter Prospective Italian Study
Brief Title: ERCP Biliary Cannulation Success Using ESGE Algorithm
Acronym: BILINCE
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Societa Italiana di Endoscopia Digestiva (Other)
Responsible Party: Principal Investigator, Alberto Mariani, Principal Investigator, IRCCS San Raffaele
Other Study IDs: BILINCE
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Biliary Tract Diseases
Keywords: ERCP; biliary cannulation; post-ERCP complications
MeSH Terms: conditions — Biliary Tract Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Papillary cannulation attempts have been shown to be an independent predictor of post-ERCP pancreatitis (PEP) when they are repeated more than 5 times or for 5 minutes or when the pancreatic duct is opacified or cannulated by using guidewire more than 1 time. In order to reduce complications, the 2016 ESGE guideline recommends a precise sequence of alternative cannulation techniques to the primary guidewire approach before exceeding the stated limits. However, there are no published data about the routinary application of this biliary cannulation algorithm.

The investigators hypothesised that the ESGE algorithm predicts an increased cannulation success. Nevertheless, it's unclear if this benefit is also associated with a decreased risk of complications, mainly post-procedural pancreatitis.

DETAILED DESCRIPTION:
Multicenter prospective observational study, which was promoted by SIED (the Italian Society of Digestive Endoscopy) involving Italian Centers that perform ERCP.

The study was approved from the Ethics Committee in 2020 with an expected enrollment of 800 patients over three years, with the potential to enroll patients for an extended period of time.

Each Center have to enroll a minimum of 15 consecutive patients, depending on the number of enrolling centers.

Each patient need to undergo ERCP by using the different cannulation techniques reported in the ESGE algorithm, which are numbered from 1 (easy cannulation) to 9 (difficult cannulation).

Digital data entry (RedCap application) are divided in three part: 1. before ERCP (patient demographics, indications for ERCP, the degree of anesthetic risk (ASA 1-3), any prophylactic therapy for pancreatitis, any assumption/interruption of anti-platelet and/or anti-coagulant drugs, the type of sedation); 2. ERCP (cannulation details according to ESGE algorithm, difficulty and duration of the procedure, final diagnosis, expertise of the endoscopist); 3. After ERCP (early and at 30-days complications, defined and graded according to the Cotton classification).

ELIGIBILITY:
Inclusion criteria:

* patients > 18 years of age;
* native papilla;
* signed Informed Consent;

Exclusion criteria:

* previous biliary sphincterotomy;
* post-surgical ERCP;
* ampulloma or papilla involved by a tumor;
* pancreatic endotherapy;
* patients unable to give consent for the procedure;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with either benign or primary/secondary malignant bile duct disease.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Success of ERCP biliary cannulation rate | At the end of the procedure.
  Success obtained with the different cannulation techniques according with the ESGE algorithm

SECONDARY OUTCOMES:
ERCP complication rates | At 0-72 hours, and at 30-days after the procedure.
  pancreatitis, bleeding, perforation, or cholangitis according with the ESGE algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Mariani, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS OSpedale San Raffaele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided